CLINICAL TRIAL: NCT02898272
Title: SCCOR Minorities Observational Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jessica Bon Field, Assistant Professor, University of Pittsburgh
Other Study IDs: PRO16040015
Record Dates: First submitted 2016-08-15; First posted 2016-09-13 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood specimens will be obtained and stored for later analysis, which may include measurement of proteins, RNA expression, DNA.
Oversight: Data Monitoring Committee: No

SUMMARY:
The SCCOR Minorities study will recruit minority participants from the COPDGene cohort, in whom the University of Pittsburgh has already obtained baseline and five year data, in order to enhance bone mineral density and vascular function data collection from minority smokers. Dual X-ray absorptiometry (DXA) scans will be obtained to measure bone mineral density. Non-invasive vascular studies will be performed to measure endothelial function. Questionnaires regarding symptoms and activity levels will be administered and a blood sample will be obtained in participants in which blood samples are not already available from the COPDGene study visits.

ELIGIBILITY:
Inclusion Criteria:

* African American male and female subjects participating in COPDGene study

Exclusion Criteria:

* caucasians
* pregnant women

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - African American male and female subjects participating in COPDGene study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Dual Xray Absorptiometry measurement of lumbar spine and hip bone mineral density. | As this is a cross-sectional collection of data, the outcome will be measured once at the first and only study visit.

SECONDARY OUTCOMES:
Measurement of carotid artery intimal thickness with ultrasound | As this is a cross-sectional collection of data, the outcome will be measured once at the first and only study visit.